CLINICAL TRIAL: NCT03959332
Title: A Phase I, Single-Centre, Open-Label, Parallel, Two Dose Level Study to Investigate the Pharmacokinetics, Safety, and Tolerability Following a Single Dose of Baloxavir Marboxil in Healthy Chinese Volunteers
Brief Title: Study to Assess the Pharmacokinetics, Safety and Tolerability of Baloxavir Marboxil in Healthy Chinese Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: YP40902
Record Dates: First submitted 2019-05-21; First posted 2019-05-22 (Actual); Results first posted 2020-06-22 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — baloxavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baloxavir Marboxil 40 mg (Experimental)
  Interventions: Drug: Baloxavir Marboxil
- Baloxavir Marboxil 80 mg (Experimental)
  Interventions: Drug: Baloxavir Marboxil

INTERVENTIONS:
Drug: Baloxavir Marboxil — Participants will receive either 40 mg or 80 mg of baloxavir marboxil on Day 1 as a single oral dose.
  Other Names: Xofluza

SUMMARY:
This study will evaluate the pharmacokinetics, safety and tolerability of a single oral dose of baloxavir marboxil (40 mg or 80 mg) in healthy Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Chinese participants must have Chinese parents and grandparents, all of whom were born in China.
* Healthy status as defined by absence of evidence of any active or chronic disease
* Participants whose body weight is ≥50 to <80 kg and body mass index is ≥18.5 to <26 kg/m2

Exclusion Criteria:

* Participants with a history of stomach, vagus nerve, or intestinal surgery (except for appendectomy)
* Participants who have a history of allergic symptoms including food allergy (Note: Non-active allergic rhinitis will be allowed)
* Participants who require chronic drug therapy or those who have used drugs within 3 days prior to screening or within 14 days prior to Day -1
* Participants who have used alcohol-containing, caffeine-containing, grapefruit containing, or St. John's wort-containing products within 72 hours prior to Day -1
* Participants who have used tobacco- or nicotine-containing products within 24 weeks prior to screening
* Participants who have donated > 400 mL of blood within 12 weeks or > 200 mL of blood within 4 weeks prior to screening, or have donated any amount of blood between screening and Day -1

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Retout S, De Buck S, Jolivet S, Duval V, Cosson V. A Pharmacokinetics-Time to Alleviation of Symptoms Model to Support Extrapolation of Baloxavir Marboxil Clinical Efficacy in Different Ethnic Groups with Influenza A or B. Clin Pharmacol Ther. 2022 Aug;112(2):372-381. doi: 10.1002/cpt.2648. Epub 2022 Jun 10. PMID 35585696
- [Derived] Liu Y, Retout S, Duval V, Jia J, Zou Y, Wang Y, Cosson V, Jolivet S, De Buck S. Pharmacokinetics, safety, and simulated efficacy of an influenza treatment, baloxavir marboxil, in Chinese individuals. Clin Transl Sci. 2022 May;15(5):1196-1203. doi: 10.1111/cts.13237. Epub 2022 Feb 19. PMID 35176206

RESULTS

PARTICIPANT FLOW:
Groups:
- Baloxavir Marboxil 40 mg; Baloxavir Marboxil 80 mg: Administered orally on Day 1
Period: Overall Study
Arm/Group | Baloxavir Marboxil 40 mg | Baloxavir Marboxil 80 mg
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baloxavir Marboxil 40 mg | Baloxavir Marboxil 80 mg | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (5.82) | 29.5 (6.09) | 28.8 (5.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 16 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 16 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Baloxavir marboxil and baloxavir concentrations were analyzed by validated Liquid Chromatography with tandem mass spectrometry (LC-MS/MS). Non-compartmental analysis was employed to estimate the PK parameters.
Time Frame: Pre-dose and at 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48,72, 120, 168, 216, 264, and 336 hours post-dose
Population: Only participants with quantifiable drug plasma concentrations were included in the parameter estimate.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Baloxavir Marboxil 40 mg | Baloxavir Marboxil 80 mg
Number analyzed (Participants) | 16 | 16
nanogram per milliliter (ng/mL)
  Baloxavir Marboxil: number analyzed (Participants) | 0 | 2
  Baloxavir Marboxil |  | 0.5133 (3.7)
  Baloxavir | 107.6 (24.2) | 206.9 (38.3)

2. Primary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Baloxavir marboxil and baloxavir concentrations were analyzed by LC-MS/MS. Non-compartmental analysis was employed to estimate the PK parameters.
Time Frame: Pre-dose and at 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48,72, 120, 168, 216, 264, and 336 hours post-dose
Population: Only participants with quantifiable drug plasma concentrations were included in the parameter estimate.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Baloxavir Marboxil 40 mg | Baloxavir Marboxil 80 mg
Number analyzed (Participants) | 16 | 16
hours (h)
  Baloxavir Marboxil: number analyzed (Participants) | 0 | 2
  Baloxavir Marboxil |  | 5.50 [5.00 to 6.00]
  Baloxavir | 4.00 [3.00 to 6.00] | 4.00 [3.00 to 5.00]

3. Primary Outcome: Area Under the Concentration to Time Curve From Time 0 to Infinity (AUC0-inf)
Description: as for outcome 2
Time Frame: Pre-dose and at 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48,72, 120, 168, 216, 264, and 336 hours post-dose
Population: Only participants with quantifiable drug plasma concentrations were included in the parameter estimate.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Baloxavir Marboxil 40 mg | Baloxavir Marboxil 80 mg
Number analyzed (Participants) | 16 | 16
ng*h/mL
  Baloxavir Marboxil: number analyzed (Participants) | 0 | 0
  Baloxavir | 6955 (25.5) | 9643 (29.4)

4. Primary Outcome: Area Under the Concentration to Time Curve From Time 0 to Last Quantifiable Concentration (AUC0-last)
Description: as for outcome 2
Time Frame: Pre-dose and at 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48,72, 120, 168, 216, 264, and 336 hours post-dose
Population: Only participants with quantifiable drug plasma concentrations were included in the parameter estimate.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Baloxavir Marboxil 40 mg | Baloxavir Marboxil 80 mg
Number analyzed (Participants) | 16 | 16
ng*h/mL
  Baloxavir Marboxil: number analyzed (Participants) | 0 | 0
  Baloxavir | 6442 (24.3) | 9218 (29.2)

5. Primary Outcome: Area Under the Concentration to Time Curve From Time 0 to Time t (AUC0-t)
Description: Time t may be chosen as a time point where evaluable concentrations are available in at least 90% of participants. Baloxavir marboxil and baloxavir concentrations were analyzed by LC-MS/MS. Non-compartmental analysis was employed to estimate the PK parameters.
Time Frame: Pre-dose and at 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48,72, 120, 168, 216, 264, and 336 hours post-dose
Population: Only participants with quantifiable drug plasma concentrations were included in the parameter estimate.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Baloxavir Marboxil 40 mg | Baloxavir Marboxil 80 mg
Number analyzed (Participants) | 16 | 16
ng*h/mL
  Baloxavir Marboxil: number analyzed (Participants) | 0 | 0
  Baloxavir | 6442 (24.3) | 9218 (29.2)

6. Primary Outcome: Terminal Elimination Half-Life (T1/2)
Description: as for outcome 2
Time Frame: Pre-dose and at 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48,72, 120, 168, 216, 264, and 336 hours post-dose
Population: Only participants with quantifiable drug plasma concentrations were included in the parameter estimate.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (h)
Arm/Group | Baloxavir Marboxil 40 mg | Baloxavir Marboxil 80 mg
Number analyzed (Participants) | 16 | 16
hours (h)
  Baloxavir Marboxil: number analyzed (Participants) | 0 | 0
  Baloxavir | 99.74 (18.0) | 88.89 (17.1)

7. Primary Outcome: Apparent Total Oral Clearance (CL/F)
Description: as for outcome 2
Time Frame: Pre-dose and at 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48,72, 120, 168, 216, 264, and 336 hours post-dose
Population: Only participants with quantifiable drug plasma concentrations were included in the parameter estimate.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)/h
Arm/Group | Baloxavir Marboxil 40 mg | Baloxavir Marboxil 80 mg
Number analyzed (Participants) | 16 | 16
Liters (L)/h
  Baloxavir Marboxil: number analyzed (Participants) | 0 | 0
  Baloxavir | 4.866 (25.5) | 7.019 (29.4)

8. Primary Outcome: Apparent Oral Volume of Distribution (Vz/F)
Description: as for outcome 2
Time Frame: Pre-dose and at 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48,72, 120, 168, 216, 264, and 336 hours post-dose
Population: Only participants with quantifiable drug plasma concentrations were included in the parameter estimate.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Baloxavir Marboxil 40 mg | Baloxavir Marboxil 80 mg
Number analyzed (Participants) | 16 | 16
L
  Baloxavir Marboxil: number analyzed (Participants) | 0 | 0
  Baloxavir | 700.1 (26.6) | 900.1 (31.4)

9. Primary Outcome: Plasma Concentrations 24 (C24), 48 (C48), and 72 Hours (C72) Postdose
Description: as for outcome 2
Time Frame: 24, 48 and 72 hours postdose
Population: Only participants with quantifiable drug plasma concentrations were included in the parameter estimate.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Baloxavir Marboxil 40 mg | Baloxavir Marboxil 80 mg
Number analyzed (Participants) | 16 | 16
ng/mL
  Baloxavir Marboxil: number analyzed (Participants) | 0 | 0
  Baloxavir C24 | 56.40 (22.8) | 92.01 (27.9)
  Baloxavir C48: number analyzed (Participants) | 16 | 14
  Baloxavir C48 | 41.38 (22.9) | 60.33 (33.2)
  Baloxavir C72 | 29.27 (25.0) | 41.78 (31.6)

10. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Time Frame: Up to Day 15
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil 40 mg | Baloxavir Marboxil 80 mg
Number analyzed (Participants) | 16 | 16
percentage of participants | 18.8 | 68.8

ADVERSE EVENTS:
Time Frame: Baseline up to Day 15
Arm/Group | Baloxavir Marboxil 40 mg | Baloxavir Marboxil 80 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 3/16 | 11/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Baloxavir Marboxil 40 mg (N=16) | Baloxavir Marboxil 80 mg (N=16)
Blood bilirubin increased (Investigations) | 1 | 2
Blood uric acid increased (Investigations) | 1 | 2
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Defect conduction intraventricular (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT03959332/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/32/NCT03959332/SAP_001.pdf